CLINICAL TRIAL: NCT02613013
Title: Laser Peripheral Iridotomy Plus Laser Peripheral Iridoplasty for Primary Angle Closure With Multi-mechanism Based on UBM: A Randomized Controlled Trial
Brief Title: Laser Peripheral Iridotomy Plus Laser Peripheral Iridoplasty for Primary Angle Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Beijing Tongren Hospital (Other); Wenzhou Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Huazhong University of Science and Technology (Other); The Third Hospital of HanDan (Other); Third Affiliated Hospital of Third Military Medical University (Other); Central South University (Other); He University (Other); Hebei Provincial Eye Hospital (Other)
Responsible Party: Principal Investigator, xiulan zhang, MD,PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015019
Record Dates: First submitted 2015-11-05; First posted 2015-11-24 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Lasers; Pilocarpine; SLC7A7 protein, human; proxymetacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single LPI (Active Comparator): LPI was performed with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA). 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia will be administered. The treatment site was selected in the superior nasal iris or in a crypt, where present. Treatment was initiated with a pulse of 3-5mJ, the power was increased until patency was achieved, the opening of iris >0.1mm. and patency was determined by direct visualization of the posterior chamber.
  Interventions: Device: neodymium:yttrium-aluminum- garnet laser; Drug: Pilocarpine; Drug: Proparacaine; Procedure: LPI
- LPIP plus LPI (Experimental): LPIP was applied with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA). 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia will be administered. Twenty to 30 spots of 250-300 mW power with 300-500 microns of size and duration of 400-500 ms were applied. Power was modified arbitrarily until an effective iris contraction was obtained. Effective iris contraction was considered as a concentric movement around the laser spot, with minimal iris pigmentation and immediate angle opening observed through the lens mirrors using a Goldmann lens. Power was lowered if there was any bursting sound perceived, pigment dispersion, air bubbles or considerable pain. LPI was performed after LPIP procedure
  Interventions: Device: neodymium:yttrium-aluminum- garnet laser; Device: frequency-doubled Q-switched neodymium:yttrium-aluminum-garnet 532-nm laser; Drug: Pilocarpine; Procedure: LPIP plus LPI; Drug: Proparacaine

INTERVENTIONS:
Device: neodymium:yttrium-aluminum- garnet laser — a neodymium:yttrium-aluminum- garnet laser was used to perform the LPI
Device: frequency-doubled Q-switched neodymium:yttrium-aluminum-garnet 532-nm laser — a frequency-doubled Q-switched neodymium:yttrium-aluminum-garnet 532-nm laser was used to perform the LPIP
  Arms: LPIP plus LPI
Drug: Pilocarpine — 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia (Proparacaine) will be administered
Procedure: LPIP plus LPI — LPIP was applied with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA). 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia will be administered. Twenty to 30 spots of 250-300 mW power with 300-500 microns of size and duration of 400-500 ms were applied. Power was modified arbitrarily until an effective iris contraction was obtained. Effective iris contraction was considered as a concentric movement around the laser spot, with minimal iris pigmentation and immediate angle opening observed through the lens mirrors using a Goldmann lens. Power was lowered if there was any bursting sound perceived, pigment dispersion, air bubbles or considerable pain. LPI was performed after LPIP procedure.
  Arms: LPIP plus LPI
Drug: Proparacaine — 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia (Proparacaine) will be administered
Procedure: LPI — LPI was performed with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA). 30 minutes prior to the procedure, a drop of 2% pilocarpine will be instilled into the eye every 15 minutes, Topical anaesthesia (Proparacaine) will be administered. The treatment site was selected in the superior nasal iris or in a crypt, where present. Treatment was initiated with a pulse of 3-5mJ, the power was increased until patency was achieved, the opening of iris >0.1mm. and patency was determined by direct visualization of the posterior chamber.
  Arms: single LPI

SUMMARY:
This is a 10-centre randomized controlled clinical trial to explore whether laser peripheral iridoplasty (LPIP) plus laser peripheral iridotomy (LPI) is more effective than single LPI to control the progression of primary angle closure with multi-mechanism based on the UBM classification.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary angle closure (PAC), with IOP≤30mmHg and PAS≤270°.
2. PAC with multi-mechanism based on UBM examination (multi-mechanism is defined as primary angle closure is caused by pupil block plus at least one kind of non-pupil block factors like (relative anterior position and thick of the ciliary body, the big volume of the iris, the anterior location of the iris insertion into the ciliary body)or any two or more kinds of combination.
3. Visual acuity≥ 20/40
4. Age between 40-75 years old Chinese people

If both eyes of a patient are eligible for the study, the e eye had worse visual acuity will be selected. Only one eye per patient is eligible for the study.

Drug washout:

Eligible patients who are already on anti-glaucoma medications are required to have drug washout before being randomized. Various medications have different washout periods: Prostaglandin analogues 4 weeks, Beta blockers 3 weeks, Adrenergic agonist 2 weeks, Cholinergic agonist 5 days, Carbonic Anhydrase Inhibitors 5 days. Patients whose IOP>30 mm Hg during this washout period will be stopped from further washout and be withdrawn from the study.

Exclusion Criteria:

1. Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits.
2. Angle closure due to secondary causes (subluxed lens, neovascular, uveitic, traumatic, post-operative)
3. Previous incisional intraocular surgery or ocular laser in study eye (LPI or LPIP, cyclodestructive procedure, cataract surgery)
4. Primary angle closure with glaucomatous neuropathy.
5. Have cataract in the studying eye and anticipated to have cataract surgery in the coming 3 years; the existing cataract affect visual field examination and fundus examination; the visual acuity <20/40 due to the existing cataract.
6. Who are using IOP lowing drugs and do not have drug washout
7. Need for glaucoma surgery combined with other ocular procedures (i.e. cataract surgery, penetrating keratoplasty, or retinal surgery) or anticipated need for urgent additional ocular surgery
8. Coexisting other ocular diseases (i.e. cornea abnormal or cornea infection, Iridocorneal endothelial syndrome or anterior segment dysgenesis, nanophthalmos, high myopia (>6.0D), Chronic or recurrent uveitis, ocular cancer, trauma, central retinal vein occlusion, central retinal artery occlusion, retinal detachment)
9. cornea endothelium counting <1000/mm2
10. need local or systemic steroid long-term use
11. Unwilling to discontinue contact lens use after surgery
12. Who are taking parting in other drug clinical trials
13. Pregnant or nursing women
14. Severe systemic disease (i.e. diabetes mellitus, hypertension, the end stage of cardiac disease, nephropathy disease, respiratory disease and cancer.
15. Allergic to pilocarpine or alcaine
16. Contraindication to ocular laser diseases.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Progression rate determined by number of patients who progress after laser treatment for each group. | 3 years
  PAC progression defined as presence of any of the following:
  1. Acute angle closure crisis
  2. Intraocular (IOP) was 8mmHg higher than initiation 1 month after the laser procedure
  3. IOP was ≥22mmHg when measured three times of continuous 1 month after the lase procedure
  4. The progression of peripheral anterior synechiae ≥ 1 clock hour within 3 years after the laser procedure as measured by gonioscopic examination.
  5. glaucomatous neuropathy within 3 years after the laser procedure

SECONDARY OUTCOMES:
Additional medication or surgery required questionnaire | 3 years
  1. the medication required to control the IOP
  2. the additional surgery required to control the progression of the PAC
The change of the best corrected visual acuity after the laser procedure | 3 years
The number of the cornea endothelial cells | 3 years
The change in angle width and configuration as measured by ultrasound biomicroscopy (UBM) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen S, Lv J, Fan S, Zhang H, Xie L, Xu L, Jiang B, Yuan H, Liang Y, Li S, Chen P, Zhang X, Wang N; Multi-mechanism Angle Closure Study (MACs) group. Laser peripheral iridotomy versus laser peripheral iridotomy plus laser peripheral iridoplasty in the treatment of multi-mechanism angle closure: study protocol for a randomized controlled trial. Trials. 2017 Mar 17;18(1):130. doi: 10.1186/s13063-017-1860-4. PMID 28302178